CLINICAL TRIAL: NCT05453916
Title: A Randomized Single-Blind Controlled Trial Comparing the Efficacy of Nitazoxanide Versus Rifaximin in Adult Patients With Irritable Bowel Syndrome Without Constipation
Brief Title: Comparing the Efficacy of Nitazoxanide Versus Rifaximin in Adult Patients With Irritable Bowel Syndrome Without Constipation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Principle Investigator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202207MH1
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — nitazoxanide; Tablets; Rifaximin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Experimental): patients receiving treatment with Nitazoxanide 500 mg two times daily for 14 days
  Interventions: Drug: Nitazoxanide 500Mg Oral Tablet
- Rifaximin (Active Comparator): patients receiving treatment rifaximin at a dose of 550 mg three times daily for 14 days.
  Interventions: Drug: Rifaximin 550Mg Tab

INTERVENTIONS:
Drug: Nitazoxanide 500Mg Oral Tablet — patients receiving treatment with Nitazoxanide 500 mg two times daily for 14 days
  Arms: Nitazoxanide
Drug: Rifaximin 550Mg Tab — patients receiving treatment rifaximin at a dose of 550 mg three times daily for 14 days
  Arms: Rifaximin

SUMMARY:
This study aim to compare the efficacy of nitazoxanide in 2-week course of treatment with rifaximin in treating diarrhea associated with IBS. We also aim to study its effect over 10 weeks after treatment to evaluate its efficacy in eradicating symptoms of IBS in the long run.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Patients suffering from diarrhea-predominant IBS according to Rome III criteria.
* Active symptoms for at least 2 weeks
* Abdominal Pain Intensity: weekly average of worst daily (in past 24 hours) abdominal pain score of > 3.0 on a 0-to-10-point scale and Stool Consistency: at least one stool with a consistency of Type 6 or Type 7 Bristol stool score (BSS) on at least 2 days per week
* Report no restriction whatsoever on their diet.

Exclusion Criteria:

* Presence of liver disease, malignancy, severe malabsorption, bedridden, endocrinological disorders, or severe chronic obstructive pulmonary disease.
* Patients who have undergone abdominal surgeries except for appendectomy and/or cholecystectomy and/or hysterectomy.
* Patients who consumed any medications that may affect bowel function within the last 2 weeks such as antibiotics, probiotics, prebiotics, antispasmodics, antidiarrheals, narcotics, or any other medication that may alter bowel function
* Patients on antidepressants or antipsychotics starting within the last six weeks before eligibility check.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects Who Had Adequate Relief of Global IBS Symptoms for at Least 2 of the 4 Weeks During the Primary Evaluation Period | 6 weeks
  The primary outcome measure is assessed during the 4-week period (ie, Weeks 3 through 6) immediately following 2 weeks of treatment with study drug

SECONDARY OUTCOMES:
Proportion of Subjects Who Had Adequate Relief of IBS-related Bloating for at Least 2 of the 4 Weeks During the Primary Evaluation Period (ie, Weeks 3 Through 6) | 6 weeks
  Proportion of Subjects Who Had Adequate Relief of IBS-related Bloating for at Least 2 of the 4 Weeks During the Primary Evaluation Period (ie, Weeks 3 Through 6)

OTHER OUTCOMES:
Biological markers | 6 weeks - 12 weeks
  The serological outcomes included the variation in interleukin-6 and anti-cdtB levels

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, University of Sadat city, Madīnat as Sādāt, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided